CLINICAL TRIAL: NCT01348451
Title: A Phase l, Open-label, First in Human, Feasibility and Safety Study of Human Spinal Cord Derived Neural Stem Cell Transplantation for the Treatment of Amyotrophic Lateral Sclerosis
Brief Title: Human Spinal Cord Derived Neural Stem Cell Transplantation for the Treatment of Amyotrophic Lateral Sclerosis
Acronym: ALS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Neuralstem Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NS2008-1
Record Dates: First submitted 2011-04-28; First posted 2011-05-05 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Human spinal cord derived neural stem cell transplantation; ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- surgery (Experimental): A sequential design of five groups will be utilized to reduce risk to subjects. The first group (Group A) will include six subjects and the subsequent groups will include three subjects per group. Each group represents both different inclusion criteria and location of surgery.
  Interventions: Device: surgical implantation

INTERVENTIONS:
Device: surgical implantation — human spinal cord stem cell implantation in ALS patients

SUMMARY:
This is a first-in-human trial of spinal derived stem cells transplanted into the spinal cord of patients with Amyotrophic Lateral Sclerosis (ALS). The goal of the study is to see if the cells and the procedure to transplant them are safe.

DETAILED DESCRIPTION:
These stem cells are called Human Spinal Stem Cells (HSSC) and have been engineered from the spinal cord of a single fetus electively aborted after 8 weeks of gestation. The tissue was obtained with the mother's consent. The cells will be transplanted into the ALS patient's spinal cord after laminectomy, an operation that removes bone surrounding the spine. After the spinal cord is exposed, a device manufactured for this purpose will be mounted onto the patient and will hold a syringe filled with the cells. The syringe will have a needle attached and the needle will enter the spinal cord in specified areas. The device will minimize trauma to the spinal cord by the needle by making the puncture precise and steady and injecting the material at a slow and steady speed.

ALS is a universally fatal neurodegenerative condition that causes weakness leading to paralysis and death. Life expectancy is 2-5 years. The cause is unknown and there is no effective treatment. Previous research has shown that on autopsy, ALS patients are found to have increased levels of the amino acid glutamate accumulated in the brain and spinal cord. This increase is thought to be caused by a decrease in the glutamate transporter which normally "cleans up" glutamate from the cells.

Because the HSSC are human in origin, their transplantation will be handled in some ways like other organ transplants in that patients will receive immunosuppressive medications to prevent the rejection of the cells. Right before and immediately after surgery patients will receive infusions of a drug called basiliximab. After surgery they will take prednisone and be tapered off that medication over one month. They will also be given two other immunosuppressive agents, tacrolimus and mycophenolate mofetil after surgery and it is expected that the patients will take these drugs for the rest of their lives.

ELIGIBILITY:
Inclusion Criteria:

1. Have the ability to understand the requirements of the study, provide written informed consent, understand and provide written authorization for the use and disclosure of Protected Health Information (PHI) [per Health Insurance Portability and Accountability Act (HIPAA) Privacy Ruling] and comply with the study procedures.
2. Subjects with sporadic or familial ALS diagnosed as laboratory-supported probable,probable or definite according to the World Federation of Neurology El Escorial Criteria (Appendix A), based on examination by the site PI.
3. Age 18 years or older.
4. Females must have a negative serum pregnancy test and practice an acceptable method of contraception or be of non-childbearing potential (post-menopausal for at least 2 years or surgically sterile [hysterectomy, oophorectomy or surgical sterilization]).
5. Geographic accessibility to the study center and the ability to travel to the clinic for study visits.
6. Presence of a willing and able caregiver.
7. Medically able to undergo lumbar or cervical laminectomy as determined by the Investigator, surgeon and anesthesiologist.
8. Medically able to tolerate immunosuppression regimen consisting of basiliximab, tacrolimus, mycophenolate mofetil, and methylprednisolone as determined by the site Investigator.
9. Agrees to the visit schedule as outlined in the informed consent.
10. Not taking riluzole (Rilutek®) or on a stable dose for ≥30 days.
11. All required vaccinations current: tetanus/diptheria (TDAP), herpes zoster/shingles(Vostavax®: within last 10 years and must be prior to surgery), pneumonia (Pneumovax®),seasonal/H1N1 flu vaccines (as appropriate for season) for Groups B-E.

Exclusion Criteria:

1. Etiology of paraplegia or weakness is due to causes other than ALS such as spinal ischemia, traumatic spinal injury, traumatic brain injury, multiple sclerosis, cerebral stroke, cerebral palsy, or infection.
2. VC < 60% predicted normal by standard nomogram at the time of screening and VC < 50% predicted normal measured supine for age at the time of surgery.
3. Current or peak Panel Reactive Antibody (PRA) due to alloantibodies > 20% receiving their first allograft.
4. Any known immunodeficiency syndrome.
5. Receipt of any investigational drug,device or biologic within 30 days of surgery.
6. Any concomitant medical disease or condition limiting the safety to participate:

   * Coagulopathy
   * Active uncontrolled infection
   * Hypotension requiring vasopressor therapy
   * Previous spinal surgery at the site of planned transplantation except for anterior cervical dissection fusion (ACDF)
   * Skin breakdown over the site of surgery
   * Malignancy (except for non-melanoma skin cancer)
   * Primary or secondary immune deficiency
   * Spinal stenosis.
7. Creatinine >1.5, liver function tests (SGOT/SGPT, Bilirubin, Alk Phos) > 2x the upper limit of normal, hematocrit/hemoglobin < 30/10, total WBC < 4000, uncontrolled hypertension (defined as systolic >180 or diastolic >100) or uncontrolled diabetes(defined as hemoglobin A1C >8), evidence of GI bleeding by hemoccult test, positive tuberculosis (TB test: PPD/Mantoux), hepatitis B or C, or human immunodeficiency virus (HIV).
8. Presence of any of the following conditions:

   * Current drug abuse or alcoholism
   * Unstable medical conditions
   * Unstable psychiatric illness including psychosis and untreated major depression within 90 days of screening
   * Positive blood test for hepatitis B or C.
9. Any condition that the site PI feels may interfere with participation in the study.
10. Any condition that the surgeon feels may pose complications for the surgery.
11. Known hypersensitivity to basiliximab, tacrolimus, mycophenolate mofetil, or methylprednisolone.
12. Inability to provide informed consent as determined by screening protocol.
13. Inadequate family or caregiver support as determined by the site PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2009-01; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The primary objective of this study is to determine the safety of human spinal cord-derived neural stem cell transplantation for the treatment of amyotrophic lateral sclerosis. | The primary outcome measure will be assessed at study visits pre and post surgery follow-up visits, for a total of 48 months.
  The primary outcome measure is the incidence of adverse events in the study population.

SECONDARY OUTCOMES:
The Secondary Objectives of the study are to evaluate spinal stem cell transplantation therapy in this patient population. | The ALSFRS-R will be administered at -3, -2 and -1 months screening/presurgery, and at 1, 3, 6, 9, 12, 18, 24, 30, 36, 42 and 48 month follow-up/post surgery visits.
  The Secondary Outcome Measures of the study are to evaluate spinal stem cell transplantation therapy in this patient population using the following 11 assessments. 1. ALSFRS-R is a self-administered ordinal rating scale questionnaire (rating 0-4 for each question, 4 is most functional, 0-48 total) of 12 functional activities. The most functional total score is 48.
The Secondary Objectives of the study are to evaluate spinal stem cell transplantation therapy in this patient population. | The quantitative muscle strength test will be administered at -3, -2, -1 months screening/presurgery and at 1, 3, 6, 9, 12, 18, 24, 30, 36, 42 and 48 month follow-up/post surgery visits.
  2. Quantitative muscle strength testing using a hand held dynamometer (HHD): Six proximal muscle groups (knee flexion and extension, hip flexion, elbow flexion and extension and shoulder flexion) and three proximal muscle groups (wrist extension, first dorsal interosseous contraction, and ankle dorsiflexion) will be tested bilaterally using the MICROFET 2 HHD.
The Secondary Objectives of the study are to evaluate spinal stem cell transplantation therapy in this patient population. | The hand grip (bilateral) will be administered at -3, -2 and -1 months screening/presurgery, and at 1, 3, 6, 9, 12, 18, 24, 30, 36, 42 and 48 month follow-up/post surgery visits.
  3. Hand grip (bilateral) will be measured using the Jaymar Grip dynamometer.
The Secondary Objectives of the study are to evaluate spinal stem cell transplantation therapy in this patient population. | The vital capacity (VC) will be measured at -3, -2 and -1 months and -7 days screening/presurgery. It will also be measured at 1, 2, 3, 6, 9, 12, 18, 24, 30, 36, 42 and 48 month follow-up/post surgery visits.
  4. Vital Capacity (VC) will be measured using the Renaissance II spirometer. Eligibility will be determined with seated and supine measurements but the secondary outcome measure will be done seated.
The Secondary Objectives of the study are to evaluate spinal stem cell transplantation therapy in this patient population. | The negative inspiratory force (NIF) will be measured at -3, -2 and -1 months and -7 days screening/presurgery. It will also be measured at 1, 2, 3, 6, 9, 12, 18, 24, 30, 36, 42 and 48 month follow-up/post surgery visits.
  5. Negative Inspiratory Force (NIF) will be measured with a Negative Inspiratory Force Gauge (Instrumentation Industries).
The Secondary Objectives of the study are to evaluate spinal stem cell transplantation therapy in this patient population. | The Electrical Impedance Myography (EIM) will be measured at -3, -2 and -1 months screening/presurgery. It will also be measured at 1, 3, 6, 9, 12, 18, 24, 30, 36, 42 and 48 month follow-up/post surgery visits.
  6. Electrical Impedance Myography (EIM) is a painless and non-invasive quantitative measure of muscle that has been shown to correlate with other physiological and semi-quantitative measures of disease progression in ALS .
The Secondary Objectives of the study are to evaluate spinal stem cell transplantation therapy in this patient population. | The comprehensive pain assessment will be performed at -3 months and -14 days screening/presurgery. It will also be performed at 2 weeks, 1, 2, 3, 6, 9, 12, 18, 24, 30, 36, 42 and 48 month follow-up/post surgery visits.
  7. Comprehensive pain assessment utilizing the Neuropathic Pain Scale (NPS).
The Secondary Objectives of the study are to evaluate spinal stem cell transplantation therapy in this patient population. | Performed during the screening and at 24 and 48 month follow-up/post surgery visits. MRI of the surgical region only, at 1, 6, 12, 18 and 36 month follow-up/post surgery visits.
  8. An MRI will be performed on the entire spine and brain with and without gadolinium contrast. An MRI of the targeted region may be performed if clinically indicated at the 2 week visit.
The Secondary Objectives of the study are to evaluate spinal stem cell transplantation therapy in this patient population. | Measurements will be taken at -3 months and -14 days at screening/presurgery and at 1, 6, 9, 12, 18, 24, 30, 36, 42 and 48 month follow-up/post surgery visits.
  9. Urodynamic parameters including incontinence and urinary retention measured by post void residual.
The Secondary Objectives of the study are to evaluate spinal stem cell transplantation therapy in this patient population. | The questionnaire will be completed at -3 months during the screening/presurgery phase and at the 3, 6, 9, 12, 18, 24, 30, 36, 42 and 48 month follow-up/post surgery visits.
  10. ALS Specific Quality of Life Questionnaire - Revised is a scale that balances physical and nonphysical factors in assessing the quality of life in ALS patients
The Secondary Objectives of the study are to evaluate spinal stem cell transplantation therapy in this patient population. | The Ashworth Spasticity Scale will be administered at -3, -2, -1 months screening/presurgery and at 1, 3, 6, 9, 12, 18, 24, 30, 36, 42 and 48 month follow-up/post surgery visits.
  11. Ashworth Spasticity Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Background] Boulis NM, Federici T, Glass JD, Lunn JS, Sakowski SA, Feldman EL. Translational stem cell therapy for amyotrophic lateral sclerosis. Nat Rev Neurol. 2011 Dec 13;8(3):172-6. doi: 10.1038/nrneurol.2011.191. PMID 22158518
- [Background] Lunn JS, Sakowski SA, Federici T, Glass JD, Boulis NM, Feldman EL. Stem cell technology for the study and treatment of motor neuron diseases. Regen Med. 2011 Mar;6(2):201-13. doi: 10.2217/rme.11.6. PMID 21391854
- [Background] Glass JD. The promise and the reality of stem-cell therapies for neurodegenerative diseases. Cerebrum. 2010 Nov;2010:24. Epub 2010 Dec 15. PMID 23447769
- [Background] Boulis N, Federici T. Surgical approach and safety of spinal cord stem cell transplantation. Neurosurgery. 2011 Feb;68(2):E599-600. doi: 10.1227/NEU.0b013e3182095e2e. No abstract available. PMID 21654562
- [Result] Glass JD, Boulis NM, Johe K, Rutkove SB, Federici T, Polak M, Kelly C, Feldman EL. Lumbar intraspinal injection of neural stem cells in patients with amyotrophic lateral sclerosis: results of a phase I trial in 12 patients. Stem Cells. 2012 Jun;30(6):1144-51. doi: 10.1002/stem.1079. PMID 22415942
- [Result] Riley J, Federici T, Polak M, Kelly C, Glass J, Raore B, Taub J, Kesner V, Feldman EL, Boulis NM. Intraspinal stem cell transplantation in amyotrophic lateral sclerosis: a phase I safety trial, technical note, and lumbar safety outcomes. Neurosurgery. 2012 Aug;71(2):405-16; discussion 416. doi: 10.1227/NEU.0b013e31825ca05f. PMID 22565043
- [Derived] Robberecht W, Philips T. The changing scene of amyotrophic lateral sclerosis. Nat Rev Neurosci. 2013 Apr;14(4):248-64. doi: 10.1038/nrn3430. Epub 2013 Mar 6. PMID 23463272
- See also: Related Info — http://neuralstem.com